CLINICAL TRIAL: NCT06955091
Title: Effects of Contrast Strength Training on Agility, Power and Explosive Speed in Badminton Players
Brief Title: Effects of Contrast Strength Training in Badminton Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RECR & AHS/24/0464
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Sports
Keywords: agility; badminton; power; resistance training; speed

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Contrast strength Training group (Experimental): 24 for contrast strength training bench press, pull over, half squat and forward lunge.
  Interventions: Other: contrast strength training
- Group B: Control Group (No Intervention): 24 Participants of the control group will follow their badminton practice and basic skills practice over the same duration with no strength training design

INTERVENTIONS:
Other: contrast strength training — For eight weeks players performed Contrast strength training included bench press, pull-over, half squat, and forward lunge. Each session began with a 10-minute warm-up (jogging, dynamic stretching, and basic weightlifting exercises) and ended with a 5-minute cool-down. Training was performed twice a week for 8 weeks on non-consecutive days (Tuesday and Thursday). Exercises were done using free weights at 40-80% of 1-repetition maximum, in 3-4 sets of 2-4 repetitions
  Arms: Group A: Contrast strength Training group

SUMMARY:
Badminton is one of the most popular sports worldwide. In general, badminton jumping actions have two goals: achieve maximum height and reach a precise location using certain body movements. Both objectives are important in badminton and must be considered when conducting practical training sessions and imparting techniques. The players should have agility to move on the court forward sideward and backward to do many actions with high speed. They require sports specific training to achieve power, stability and agility in the ground for a powerful performance. Contrast strength training is multi-intervention programs and it has a certain influence on agility, power and speed. A sample size of 48 badminton players from Pakistan Sports Board, university level and badminton club players will be taken through Non-Probability Convenience Sampling technique. Sample size of players with age group between 17-28 years will be taken. Players will be selected on the basis of inclusion and exclusion criteria and will be equally divided into two groups by random number generator table. Group A experimental group will perform contrast strength training. Group B participants of the control group will follow their standard badminton practice over the same duration with no strength training design. Before and after completion of the respective training agility and power will be assessed through t-test and vertical jump test. For explosive speed 40-yard dash will be performed. Data will be analyzed by using Statistical Package for the Social Sciences (SPSS) for Windows Version 25.

DETAILED DESCRIPTION:
This study aims to examine the effects of contrast strength training on agility, power, and speed in badminton players. Data will be analyzed using the Statistical Package for the Social Sciences (SPSS), version 25

ELIGIBILITY:
Inclusion Criteria:

* • Both male and female athletes.

  * Participants between the age of 17-28.(10)
  * Have been playing on a regular basis three-four times a week(21)
  * Players must have been playing badminton for more than 2 years.(22)

Exclusion Criteria:

* Athletes with systemic and neuromuscular issue(1)
* Players have musculoskeletal problem which can hinder the trainings.(10)
* Received surgery in the three years prior to the study or had undergone rehabilitation within the past year.(1)
* Could not commit to full participation in the study's training regimes.
* Did not practice any training in the last six months(10)
* History of injury in past 6 months(10)
* Previous history of fracture, previous injury, open wounds.(10)

Ages: 17 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Agility T Test | 8 weeks
  The T-test, an accurate approach with a good intra-trial reliability score was used to measure agility. The participants were told to touch the first cone with their right hand after running 9.14 meters from the starting line. They shuffled to the second cone, which was 4.57 meters to the left, then to the third, which was 9.14 meters to the right, touching it with their right hand, then reversing to the starting line after shuffling 4.57 meters to the center cone and touching it with their left
Vertical Jump Power Test | 8 weeks
  The participant applies chalk to the tips of their fingers. After standing away from the wall, the individual uses both arms and legs to help project their body upwards and jumped as high as they are capable of. Attempt to touch the wall at the top of the jump. Power will be measured by Sargent Test.
40-Yd Speed Test | 8 weeks
  Speed was evaluated using the 40-Yard Sprint Test, which involves completing a single maximum-effort sprint over a 40-yard distance while recording the time. The purpose of this test was to assess the participants' 40-yard sprint performance.

CONTACTS AND LOCATIONS:
Overall Officials: Muzna ShahidMunir, Principal Investigator — Riphah International University
Locations (1):
- Pakistan sports Board Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maio Alves JM, Rebelo AN, Abrantes C, Sampaio J. Short-term effects of complex and contrast training in soccer players' vertical jump, sprint, and agility abilities. J Strength Cond Res. 2010 Apr;24(4):936-41. doi: 10.1519/JSC.0b013e3181c7c5fd. PMID 20300035
- [Background] Wisloff U, Castagna C, Helgerud J, Jones R, Hoff J. Strong correlation of maximal squat strength with sprint performance and vertical jump height in elite soccer players. Br J Sports Med. 2004 Jun;38(3):285-8. doi: 10.1136/bjsm.2002.002071. PMID 15155427
- [Background] Malwanage KT, Senadheera VV, Dassanayake TL. Effect of balance training on footwork performance in badminton: An interventional study. PLoS One. 2022 Nov 17;17(11):e0277775. doi: 10.1371/journal.pone.0277775. eCollection 2022. PMID 36395192
- [Background] Chandra S, Sharma A, Malhotra N, Rizvi MR, Kumari S. Effects of Plyometric Training on the Agility, Speed, and Explosive Power of Male Collegiate Badminton Players. J Lifestyle Med. 2023 Feb 28;13(1):52-58. doi: 10.15280/jlm.2023.13.1.52. PMID 37250280